CLINICAL TRIAL: NCT01619254
Title: Hand Hygiene Promotion Activities: Effect on Intestinal Parasitic Infections and Anaemia Among School-aged Children in Eastern Tigray, Ethiopia: a Factorial Randomised Controlled Trial
Brief Title: Impact of Hand Hygiene Activities on the Prevention of Intestinal Parasitic Infections and Anaemia Among School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mekelle University (Other)
Collaborators: University of Alcala (Other); Maastricht University (Other)
Responsible Party: Principal Investigator, Mahmud Abdulkader, PhD fellow and Instructor, Mekelle University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: AECID
Record Dates: First submitted 2012-06-09; First posted 2012-06-14 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Intestinal Parasitic Infections; Anaemia
Keywords: Intestinal parasitic infections; Anaemia; School-aged children; Hand washing and nail clipping
MeSH Terms: conditions — Anemia | interventions — Hand Disinfection; Soaps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Hand hygiene (Experimental): Hand washing with soap measures will be carried out as an intervention activity
  Interventions: Behavioral: Hand washing with soap and hand finger nail clipping
- Hand finger nail hygiene (Experimental): Hand finger nail clipping activities
  Interventions: Behavioral: Hand washing with soap and hand finger nail clipping
- Hand and finger nails hygiene (Experimental): Both hand washing with soap and hand finger nail clipping activities will be implemented
  Interventions: Behavioral: Hand washing with soap and hand finger nail clipping
- Customary practice (Placebo Comparator): No hand washing with soap and nail clipping activities. House holds and children assigned to the control group will not have the interventions (hand washing with soap and nail clipping activities)
  Interventions: Behavioral: Hand washing with soap and hand finger nail clipping

INTERVENTIONS:
Behavioral: Hand washing with soap and hand finger nail clipping — Assess the impact of hand washing with soap and nail clipping on child health
  Other Names: Hand washing and finger nails clipping

SUMMARY:
Impact exerted by intestinal parasitic infections is much higher in developing countries. School-aged children are at higher risk from the burden of disease, because they specially have many parasitic infections. The poor health results in deficits in physical and cognitive development and educational achievements. Nowadays, there is huge commitment among the global community to control intestinal parasitic infections and to improve nutritional status of young children in developing countries.

Large-scale anthelminthic drug administration through vertical control programmes is still required for the foreseeable future and is, therefore, recommended by the World Health Organization (WHO). However, due to the inevitability of re-infection in endemic areas, children need to be treated regularly, and once morbidity control is consolidated, the strategy must shift to transmission control emphasising access to clean water and adequate sanitation. To lower dependency on 'drug only' approach and to enhance sustainability, from the onset of control activities, complementary measures should be implemented, that depend on available resources.

Therefore, the investigators are proposing to undertake a randomised controlled trial to assess the impact of simple and easy-to-do hand hygiene intervention packages (hand washing with soap and hand finger nail clipping) on intestinal parasitic infection prevalence, intensity and re-infection rates and on haemoglobin concentration and anaemia prevalence rates among 6-15 years old schoolchildren. Our results will provide solid evidence on if and how hand hygiene practice affects infection prevalence and re-infection rates, as well as, anaemia prevalence among the highly vulnerable age group.

DETAILED DESCRIPTION:
The controlled prospective cohort study will be carried out in Kilte awlaelo wereda, north Ethiopia. A total of 216 households with at least one school-aged child (aged 6-15) will be randomly selected by systematic random sampling method. Different intervention packages will be randomised among households. Intervention activities will be implemented at household level, using the selected child within the household as study unit.

If there are more than one child per randomised household all children will receive the intervention, but only two children, selected by simple random selection method, will be included in the trial. Selected children will be screened for intestinal parasitosis, following acquisition of signed informed consent, and will be recruited for the study after treatment.

Parasite negative children in the respective households will be randomly allocated into intervention and control groups. Sequence allocation will be done in a central office by an individual who do not know and have no contact with the study sites and households.

Each intervention and control group will have a fixed number of participants, and will be subjected to only one of the study interventions. Children and households in each group will be followed-up for 6 months by trained fieldworkers and the investigators according to a developed protocol throughout the study period. Parasitological, haemoglobin and anthropometric data will be collected at entry and after six months.

ELIGIBILITY:
Inclusion Criteria:

* households and children who will give a written consent to participate in the study
* households and children who are going to stay in the area throughout the study period
* children aged 6 to 15

Exclusion Criteria:

* households and children who able to produce a written consent
* children who are under treatment
* children with age less than 6 and greater than 15 years

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 365 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
- Proportion of intestinal parasitic re-infection rates among intervention and control groups | six months
  Impact of hand hygiene activities (as intervention measures) on intestinal parasitic re-infection prevalence will be assessed.
- Proportion of intestinal parasite load (mean eggs per gram) among intervention and control groups | six months
  Impact of hand hygiene activities (as intervention measures) on intestinal parasitic infection intensity will be assessed.

SECONDARY OUTCOMES:
Proportion of anaemia prevalence rates among intervention and control groups | six months
  Impact of hand hygiene activities on the reduction of anaemia prevalence among the children will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Mahmud Ab Mahmud, PhD fellow, Principal Investigator — College of Health Scieneces, Mekelle University; Roman B Velasco, MD, PhD, Study Director — Alcala University, Madrid, Spain; Mark Spigt, MSC, PhD, Study Chair — Maastricht University, The Netherlands; Afework M Bezabeh, MSC, PhD, Study Chair — College of Health Sciences, Mekelle University; Geert J Dinant, Professor, Study Chair — Maastricht University, The Netherlands
Locations (1):
- College of Health Sciences, Mekelle University, Mek'ele, Tigray, Ethiopia

REFERENCES:
- [Derived] Mahmud MA, Spigt M, Bezabih AM, Dinant GJ, Velasco RB. Associations between intestinal parasitic infections, anaemia, and diarrhoea among school aged children, and the impact of hand-washing and nail clipping. BMC Res Notes. 2020 Jan 2;13(1):1. doi: 10.1186/s13104-019-4871-2. PMID 31898526